CLINICAL TRIAL: NCT01243866
Title: Effect of Dental Treatment on Children's Growth
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: King Fahad Armed Forces Hospital (Other Government)
Responsible Party: Dr Hiba Alkarimi, King Fahad Armed Forces Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD109
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2008-01

CONDITIONS: Dental Decay
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early treatment (Experimental): comprehensive dental treatment
  Interventions: Other: comprehensive dental treatment
- Regualr treatment (No Intervention): Regular treatment consisted of children who would be on a waiting list for regular dental treatment at KFAFH for at least 8 months
  Interventions: Other: Only emergency dental treatment

INTERVENTIONS:
Other: comprehensive dental treatment — Early treatment children were scheduled for comprehensive dental treatment over a 2-month period (from May to June 2007). All test children had their last dental treatment visit within the last 2 weeks of the second treatment month. The follow-up survey was scheduled for each child to be approximately 6-month after their dental last visit. This step was very important to make sure that all children were examined at exactly the same interval between end of treatment and when re-examined at the follow-up examination.
  Arms: Early treatment
Other: Only emergency dental treatment — Regular treatment did not receive any dental treatment in the period when the early children were treated unless they had toothache or dental infection. In that case they were treated for the pain but did not have comprehensive dental treatment
  Arms: Regualr treatment

SUMMARY:
Severe dental decay affects children physically, emotionally, socially and thereby impacts on their quality of life. Evidence from developed countries showed that children with severe dental decay weighed less than their peers and following dental treatment children's growth and quality of life improved. This suggests that treatment of severe dental decay may enhance growth and wellbeing. A study was carried out in Saudi to test that hypothesis.

ELIGIBILITY:
Inclusion Criteria:

Having dental caries with at least 2 teeth with pulpal involvement.

Exclusion Criteria:

1. Children with illness known to adversely affect growth.
2. Children who required urgent dental treatment.
3. Children on regular nutritional supplements.
4. Anaemic children with Hb levels lower than 11.0 g/dl

Ages: 72 Months to 95 Months | Sex: All
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2007-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Children's height and weight (HAZ,WAZ and BAZ) | 6 months
  children's height and weight were measured pre and 6 months post dental treatment.

SECONDARY OUTCOMES:
Quality of life (pain, sepsis, satisfaction and appetite) | 6 months
  specific general and oral quality of life health measures were examined before and after dental treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hiba A Alkarimi, PhD, Study Director — KFAFH

REFERENCES:
- [Derived] Alkarimi HA, Watt RG, Pikhart H, Jawadi AH, Sheiham A, Tsakos G. Impact of treating dental caries on schoolchildren's anthropometric, dental, satisfaction and appetite outcomes: a randomized controlled trial. BMC Public Health. 2012 Aug 29;12:706. doi: 10.1186/1471-2458-12-706. PMID 22928903